CLINICAL TRIAL: NCT01666353
Title: PET Quantitative Assessments of Solid Tumor Response to Immune Checkpoint Blockade Therapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Melanoma Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J1208; NA_00049919 (Other: JHMIRB)
Record Dates: First submitted 2012-05-18; First posted 2012-08-16 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Melanoma; Renal Cell Carcinoma (RCC); Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic response for solid tumors (Experimental): Adult patients, with documented metastatic melanoma, RCC or NSCLC, about to initiate any line of immune checkpoint blockade therapy will receive a FDG PET scan during mid treatment to check for change in disease.
  Interventions: Radiation: PET/CT imaging with [18F] 2-deoxy-2-(18F)fluoro-D-glucose (FDG)

INTERVENTIONS:
Radiation: PET/CT imaging with [18F] 2-deoxy-2-(18F)fluoro-D-glucose (FDG) — PET/CT imaging with [18F] 2-deoxy-2-(18F)fluoro-D-glucose (FDG) is a potent diagnostic tool and is able to detect melanomas and other tumors, some of which are undetectable by CT.

SUMMARY:
This study aims to develop methods for quantitative imaging of solid tumors in patients who are receiving immunotherapies that have a delayed mechanism of action.

PET imaging with [18F] 2-deoxy-2-(18F)fluoro-D-glucose (FDG) is a potent diagnostic tool and is able to detect melanomas and other tumors, some of which are undetectable by CT. FDG PET is now used commonly in detecting melanoma in humans as melanomas quite consistently have high glucose metabolism. PET with FDG can image the response of tumors to therapy, but has not been extensively evaluated in melanoma nor in immunotherapy for melanoma. PET has been shown to be highly predictive of outcomes of patients following radioimmunotherapy of lymphoma, and has shown changes in tumor glycolysis as early as 7 days after immunotherapy initiation.

In order to develop PET/CT as a tool to detect early evidence of response in patients with solid tumors receiving immune checkpoint blockade, investigators propose to perform PET/CT imaging prior to therapy, again between days 21 and 28, and finally at 4 months post-treatment initiation. Each scan will be assessed qualitatively and quantitatively. Investigators will use the PERCIST criteria to determine peak and maximum standardized uptake values corrected for lean body mass (SUL) in tumor, tumor volumes, and tumor total glycolytic volumes, and will use CT from PET/CT to measure tumor size by immune RECIST criteria. (See section on Outcome Evaluation below.) Investigators will assess whether early changes in tumor metabolism seen on FDG PET are predictive of progression free and overall survival outcomes. Through these systematic pilot studies, investigators hope to better link FDG PET measurements to individual patient responses to immune checkpoint blockade therapy and better understand and refine this emerging and often effective therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Any subject with documented metastatic melanoma, RCC or NSCLC.
3. Subjects must be scheduled to receive therapy, or received only one dose, with an anti-neoplastic agent that works by immune checkpoint blockade such as ipilimumab/Yervoy (anti-CTLA-4), MDX-1106/BMS-936558 (anti-PD-1) or MDX-1105/BMS-936559 (anti-B7-H1) mAbs.
4. Subjects must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as >10 mm with spiral CT scan.

Exclusion Criteria:

1. Patient is unable to provide informed consent
2. Patient is pregnant
3. Patient enrollment on research protocol which includes an additional mid-therapy investigational FDG PET/CT at approximately month from start of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04-16 (Actual); Primary Completion 2014-06-02 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Compare FDG PET-based qualitative and quantitative tumor response assessment with standard CT immune RECIST criteria | 6 months after completion of standard of care treatment
  To compare FDG PET-based qualitative and quantitative tumor response assessment with standard CT immune RECIST criteria in patients receiving immune checkpoint blockade therapy for melanoma, renal cell carcinoma (RCC), and non-small cell lung cancer (NSCLC). Patients will receive 2 standard of care treatment FDG scans, the first scan at the beginning of treatment and the second scan at the end of treatment. The research scan will be done between the first and second scan.

SECONDARY OUTCOMES:
Assess the use of FDG PET as a non-invasive imaging method to detect early evidence of organ inflammation in patients receiving immune checkpoint blockade therapy | 6 months after completion of standard of care treatment
  To compare FDG PET-derived SUV-based tumor metabolic activity in patients with prolonged stable partial responses to immune checkpoint blockade

CONTACTS AND LOCATIONS:
Overall Officials: Evan Lipson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Cho SY, Lipson EJ, Im HJ, Rowe SP, Gonzalez EM, Blackford A, Chirindel A, Pardoll DM, Topalian SL, Wahl RL. Prediction of Response to Immune Checkpoint Inhibitor Therapy Using Early-Time-Point 18F-FDG PET/CT Imaging in Patients with Advanced Melanoma. J Nucl Med. 2017 Sep;58(9):1421-1428. doi: 10.2967/jnumed.116.188839. Epub 2017 Mar 30. PMID 28360208